CLINICAL TRIAL: NCT06679803
Title: PA-ChatS: Feasibility of Delivering a First-Line Physical Activity Intervention After Stroke
Brief Title: Feasibility of a First-Line Physical Activity Intervention After Stroke
Acronym: PA-ChatS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIN-2024-33389; UM1TR004405 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Ischemic Stroke; Hemorrhagic Stroke
Keywords: physical activity; occupational therapy; behavioral intervention; stroke rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PA-ChatS Intervention (Experimental): Participants will receive 6, 20-30 minute intervention sessions delivered over the telephone by an occupational therapist over 6 weeks (1 session/week). They will also complete self-monitoring of step counts using a Fitbit Inspire.
  Interventions: Behavioral: Physical Activity Chats after Stroke (PA-ChatS)

INTERVENTIONS:
Behavioral: Physical Activity Chats after Stroke (PA-ChatS) — PA-ChatS consists of (1) self-monitoring step count using a Fitbit Inspire, and (2) behavioral activation for stepping activity delivered via the telephone and guided by the PA-ChatS workbook.
  Participants will receive education regarding the physical activity after stroke, American Heart/Stroke Association guidelines for post-stroke physical activity levels, and an overview of the intervention activities. They will then use the Fitbit data to monitor average daily step counts, set a new step count goals (increasing by 5 to 10% of the daily average step count from the prior week), and create a specific plan for achieving the new step count goal. The interventionist will collaboratively problem solve with the participant to identify strategies to overcome barriers to stepping activity and maintain safety.

SUMMARY:
The goal of this study is to explore a new intervention that supports physical activity within the first 6 weeks after stroke. All participants will complete assessments at weeks 0 and 7. During weeks 1 through 6, participants will use a Fitbit Inspire to track their step counts and meet with an occupational therapist one time per week. They will also complete weekly surveys. Physical activity levels will be measured using surveys and a wearable activPAL monitor 6 times during the study: Weeks 1, 3, 5, 7, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis confirmed by imaging
* Admitted to Fairview Health System (Minnesota) at the time of study enrollment or discharged to a community-based setting from Fairview Health System within 3 months before study enrollment
* Able and willing to participate fully in the study and provide informed consent or proxy consent with participant assent

Exclusion Criteria:

* Discharge anticipated to a transitional care unit, skilled nursing facility, or other non-community-based care setting
* Severe cognitive or communication impairments (inability to respond accurately to complete study screening questions or to provide informed consent or assent
* Comorbid neurological disorder (Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, myasthenia gravis, dementia, Alzheimer's disease, Huntington's disease, glioblastoma, spinal cord injury, cerebral palsy)
* Comorbid cancer, currently undergoing chemotherapy or radiation treatment
* Received inpatient treatment or was hospitalized for psychiatric condition and/or alcohol or substance abuse within the past 12 months
* Current diagnosis of a terimnal illness and/or receiving hospice care
* History of allergic reaction to adhesives that precludes the use of an adhesive necessary for adherence to activPAL measurement
* Inability to speak, read, or understand English
* Concurrent participation in another rehabilitation intervention research study
* Resides more than 50 miles outside of the Twin Cities metropolitan area
* Investigator discretion for safety or adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to PA-ChatS sessions | 6-weeks
  Percentage of participants who complete 6 out of 6 (100%) of PA-ChatS sessions. Session completion will be documented by the study intervention therapist and total count of sessions completed will be computed after the last intervention session is delivered.
Adherence to wearable activity tracker | 6-weeks
  Percentage of participants who use the wearable activity tracker (Fitbit Inspire 3) an average of 5 of 7 days/week during the 6-week intervention period. Data will be exported from Fitbit to compute average number of days per week the Fitbit was used.

SECONDARY OUTCOMES:
Acceptability of PA-ChatS Intervention | Week 7
  The Client Satisfaction Questionnaire-8 will be used to measure acceptability of the intervention. This is an 8-item measure with each item rated on a 1 to 4-point Likert-type scale, and then averaged across all 8 items. A mean score of 3 or more indicates that the intervention is generally acceptable.
Safety of the PA-ChatS intervention | Week 7
  All participants will be queried regarding possible adverse events during the study at one time-point using an adverse events questionnaire previously administered in physical activity studies after stroke.
Change in step count | Weeks 1 to 12
  The activPAL micro4 will be used to measure step count, following a 24-hour, 7-day wear protocol.
Change in sedentary time | Weeks 1 to 12
  The activPAL micro4 will be used to measure sedentary time, following a 24-hour, 7-day wear protocol. Participants will complete a daily diary indicating the sleep time. Sleep will be removed following a diary-informed method.
Adherence to step count | Week 24
  The activPAL micro4 (24/7 wear protocol) will used to measure step count. The proportion of participants achieving 7500 or more steps per day will be reported.
Adherence to sedentary time | Week 24
  The activPAL micro4 (24/7 wear protocol) will used to measure sedentary time. Participants will complete a diary to indicate sleep time, and sleep will be removed following a diary-informed method. The proportion of participants achieving 7 hours or less of sedentary time per day will be reported.
Adherence to moderate-to-vigorous physical activity | Week 24
  The International Physical Activity Questionnaire will used to measure minutes per week of moderate-to vigorous-physical activity (MVPA). The proportion of participants achieving 90 minutes or more/week of MVPA will be reported.
Adherence to strength training | Week 24
  The Muscle-Strengthening Exercise Questionnaire Short Form will used to measure days per week of strength training. The proportion of participants achieving 2 or more days per week of strength training will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kringle, PhD, OTR/L, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data related to demographics, medical and stroke history, cognitive function, mobility, self-reported psychosocial and social support measures, and physical activity data may be requested.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data and supporting documents will be made available upon reasonable request after the main results are published in a peer-reviewed journal.
Access Criteria: Requests for data sharing may be directed to the Principal Investigator. Deidentified IPD and supporting will be provided upon reasonable request through appropriate channels (Data Use Agreement).